CLINICAL TRIAL: NCT04979988
Title: Retrospective, Multicenter, Observational Study to Evaluate Clinical Real World Outcomes of Lorlatinib After Alectinib in ALK-Positive NSCLC Japanese Patients
Brief Title: Study to Evaluate Clinical Real World Outcomes of Lorlatinib After Alectinib in ALK-Positive NSCLC Japanese Patients
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B7461038
Record Dates: First submitted 2021-07-19; First posted 2021-07-28 (Actual); Results first posted 2024-04-05 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2023-10

CONDITIONS: ALK-positive Non-small-cell Lung Cancer
Keywords: ALK; Lorlatinib; Alectinib; Real World; retrospective

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Japanese patients with ALK+ NSCLC who received lorlatinib: lorlatinib as the second-line or later therapy after failure of alectinib treatment as the firstline therapy
  Interventions: Drug: Lortlatinib

INTERVENTIONS:
Drug: Lortlatinib — as provided in real world practice

SUMMARY:
To evaluate the clinical real world outcomes of lorlatinib in second/later line setting anaplastic lymphoma kinase (ALK) tyrosine kinase inhibitor (TKI) to TKI sequence sequence treatment after failure of alectinib as a first-line treatment in Japanese ALK positive non-small cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
This study is a post-approval, company-sponsored, observational study. This study is a multicenter, non-interventional, retrospective, chart review of patients with ALK+ NSCLC patients treated using lorlatinib as the second/later line therapy in Japan after failure of alectinib treatment as the first line therapy from 20 November 2018.

All decisions regarding clinical management and treatment of the participating patients were made by an investigator as part of standard care in real-world clinical setting and were not contingent upon the patient's participation in the study. Data will be collected if available per study site. Patients in this study are those who started treatment with lorlatinib from 1 May 2019 to 31 December, 2020 in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed NSCLC, with any tumor, node and metastasis (TNM) stage.
* Confirmed ALK gene rearrangement by any validated test.
* Confirmed the treatment with alectinib in the first line setting as systemic therapy in the medical record.
* Confirmed the start treatment with lorlatinib as the second/later-line therapy from 1st May 2019 to 31st December 2020.

Exclusion Criteria:

-Participating on any clinical trials of which final results has not yet been reported during the study period.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ALK-positive lung cancer diagnosed and confirmed in the medical record as receiving alectinib in the 1st line and lorlatinib in the 2nd line or later between May 2019 and December 2020.
Sampling Method: Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2021-08-02 (Actual); Primary Completion 2021-12-09 (Actual); Study Completion 2021-12-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (16):
- Japan (16):
  - Aichi Cancer Center Hospital, Nagoya, Aichi-ken
  - Fujita Health University Hospital, Toyoake, Aichi-ken
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - Kurashiki Central Hospital, Kurashiki, Okayama-ken
  - Kansai Medical University Hirakata Hospital, Hirakata, Osaka
  - Osaka International Cancer Institute, Osaka, Osaka
  - National Hospital Organization Kinki-Chuo Chest Medical Center, Sakai-shi, Osaka
  - Kinki University Hospital, Sayama, Osaka
  - Shizuoka Cancer Center, Sunto-gun, Shizuoka
  - Jichi Medical University Hospital, Shimotsuke, Tochigi
  - Juntendo University Hospital, Bunkyo-ku, Tokyo
  - National Hospital Organization Iwakuni Clinical Center, Iwakuni, Yamaguchi
  - National Hospital Organization, Yamaguchi-Ube Medical Center, Ube, Yamaguchi
  - The Cancer Institute Hospital of JFCR, Koto-ku, Tokyo
  - National Cancer Center, Tokyo
  - Toyama Prefectural Central Hospital, Toyama

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7461038

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with anaplastic lymphoma kinase (ALK) positive (+) non-small cell lung cancer (NSCLC) who started treatment with lorlatinib as the second line (2L) or later line therapy from 01-May-2019 to 31-Dec-2020 in real world clinical practice after failure of alectinib treatment as the first line therapy were observed in this retrospective chart review study. The study was conducted in Japan.
Pre-assignment Details: Data from participants were observed from start of alectinib treatment until 15-Oct-2021 (data cut-off date). Data was collected from medical records and evaluated over approximately 4 months (02-Aug-2021 to 09-Dec-2021) of this retrospective study.
Groups:
- Lorlatinib 2L: Participants with ALK+ NSCLC who started treatment with lorlatinib as the second-line therapy from 01-May-2019 to 31-Dec-2020 in real world clinical practice after failure of alectinib treatment as the first line therapy were observed in this retrospective study.
- Lorlatinib 3L or Later: Participants with ALK positive NSCLC who started treatment with lorlatinib as the third line (3L) or later line therapy from 01-May- 2019 to 31-Dec-2020 in real world clinical practice after failure of alectinib treatment as the first line therapy were observed in this retrospective study.
Period: Overall Study
Arm/Group | Lorlatinib 2L | Lorlatinib 3L or Later
Started | 29 | 22
Completed | 29 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) comprised of participants with confirmed ALK+ NSCLC who started treatment with lorlatinib as the second-line or later therapy from 01-May-2019 to 31-Dec-2020 and had confirmed treatment with alectinib in the first line setting in a medical record.
Groups:
- Total: Total of all reporting groups
Arm/Group | Lorlatinib 2L | Lorlatinib 3L or Later | Total
Number analyzed (Participants) | 29 | 22 | 51
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.2 (11.5) | 55.6 (14.8) | 55.9 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 15 | 24
  Male | 20 | 7 | 27
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Age at Start of Lorlatinib Treatment
Description: Age at start of lorlatinib treatment was entered based on the data in medical chart. If there were no details about the applicable age, the age was calculated from the date of birth to the start date of lorlatinib treatment.
Time Frame: At initiation of lorlatinib treatment, anytime between 01-May-2019 to 31-Dec-2020 (approximately 20 months); retrospective data was retrieved and analyzed during 4 months of this observational study
Population: FAS comprised of participants with confirmed ALK+ NSCLC who started treatment with lorlatinib as the second-line or later therapy from 01-May-2019 to 31-Dec-2020 and had confirmed treatment with alectinib in the first line setting in a medical record.
Measure: Mean (Standard Deviation); unit: Years
Arm/Group | Lorlatinib 2L | Lorlatinib 3L or Later
Number analyzed (Participants) | 29 | 22
Years | 57.7 (11.7) | 58.1 (14.5)

2. Primary Outcome: Height at Start of Alectinib Treatment
Time Frame: At initiation of alectinib treatment (baseline); retrospective data was retrieved and analyzed during 4 months of this observational study
Population: FAS comprised of participants with confirmed ALK+ NSCLC who started treatment with lorlatinib as the second-line or later therapy from 01-May-2019 to 31-Dec-2020 and had confirmed treatment with alectinib in the first line setting in a medical record. Here, 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Centimeter
Arm/Group | Lorlatinib 2L | Lorlatinib 3L or Later
Number analyzed (Participants) | 21 | 15
Centimeter | 165.44 (7.16) | 160.40 (9.23)

3. Primary Outcome: Height at Start of Lorlatinib Treatment
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Centimeter
Arm/Group | Lorlatinib 2L | Lorlatinib 3L or Later
Number analyzed (Participants) | 9 | 13
Centimeter | 163.16 (7.51) | 159.01 (8.81)

4. Primary Outcome: Weight at Start of Alectinib Treatment
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Lorlatinib 2L | Lorlatinib 3L or Later
Number analyzed (Participants) | 22 | 15
Kilograms | 60.52 (16.45) | 58.27 (11.83)

5. Primary Outcome: Weight at Start of Lorlatinib Treatment
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Lorlatinib 2L | Lorlatinib 3L or Later
Number analyzed (Participants) | 12 | 15
Kilograms | 61.92 (15.05) | 58.19 (14.19)

6. Primary Outcome: Body Mass Index (BMI) at Start of Alectinib Treatment
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Kilograms per meter square
Arm/Group | Lorlatinib 2L | Lorlatinib 3L or Later
Number analyzed (Participants) | 21 | 15
Kilograms per meter square | 22.10 (4.72) | 22.55 (3.77)

7. Primary Outcome: BMI at Start of Lorlatinib Treatment
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Kilograms per meter square
Arm/Group | Lorlatinib 2L | Lorlatinib 3L or Later
Number analyzed (Participants) | 9 | 13
Kilograms per meter square | 22.93 (4.74) | 22.42 (4.98)

8. Primary Outcome: Number of Participants According to Eastern Cooperative Oncology Group Performance Status (ECOG PS) at Start of Alectinib Treatment
Description: ECOG PS is used to measure quality of life of participants with grades ranging from 0 to 5; where Grade 0: fully active; Grade 1: restricted in physically strenuous activity but ambulatory; Grade 2: ambulatory and capable of all self-care but unable to carry out any work activities; Grade 3: capable of only limited self-care; Grade 4: completely disabled and Grade 5: dead. Higher scores indicated worsening of quality of life. Number of participants according to ECOG PS were presented. Participants whose ECOG PS was not known were reported under category "Unknown".
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Lorlatinib 2L | Lorlatinib 3L or Later
Number analyzed (Participants) | 29 | 22
Participants
  0 | 4 | 4
  1 | 12 | 8
  2 | 5 | 2
  3 | 1 | 2
  4 | 1 | 0
  5 | 0 | 0
  Unknown | 6 | 6

9. Primary Outcome: Number of Participants According to ECOG PS at Start of Lorlatinib Treatment
Description: as for outcome 8
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Lorlatinib 2L | Lorlatinib 3L or Later
Number analyzed (Participants) | 29 | 22
Participants
  0 | 5 | 2
  1 | 14 | 11
  2 | 3 | 2
  3 | 1 | 2
  4 | 0 | 0
  5 | 0 | 0
  Unknown | 6 | 5

10. Primary Outcome: Number of Participants According to NSCLC Histopathological Subtype
Description: Number of participants according to NSCLC histopathological subtype (adenocarcinoma, squamous cell carcinoma and adenosquamous epithelial carcinoma) were reported in this outcome measure.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Lorlatinib 2L | Lorlatinib 3L or Later
Number analyzed (Participants) | 29 | 22
Participants
  Adenocarcinoma | 27 | 21
  Squamous cell carcinoma | 1 | 1
  Adenosquamous epithelial carcinoma | 1 | 0

11. Primary Outcome: Number of Participants According to Presence of Metastases at Start of Alectinib Treatment
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Lorlatinib 2L | Lorlatinib 3L or Later
Number analyzed (Participants) | 29 | 22
Participants
  No | 0 | 0
  Yes | 28 | 22
  Unknown or unconfirmed | 1 | 0

12. Primary Outcome: Number of Participants According to Presence of Metastases at Start of Lorlatinib Treatment
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Lorlatinib 2L | Lorlatinib 3L or Later
Number analyzed (Participants) | 29 | 22
Participants
  No | 0 | 0
  Yes | 29 | 22
  Unknown or unconfirmed | 0 | 0

13. Primary Outcome: Number of Participants According to Sites of Metastases at Start of Alectinib Treatment
Description: Number of participants according to sites of metastasis at start of alectinib treatment were presented in this outcome measure. One participant could have more than one site of metastases.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Lorlatinib 2L | Lorlatinib 3L or Later
Number analyzed (Participants) | 28 | 22
Participants
  Ipsilateral lung | 9 | 9
  Contralateral lung | 5 | 7
  Lymph node affiliation | 23 | 21
  Remote lymph node | 5 | 7
  Liver | 4 | 6
  Bone | 12 | 12
  Brain | 7 | 7
  Adrenal glands | 1 | 1
  Kidney | 1 | 0
  Other | 11 | 7

14. Primary Outcome: Number of Participants According to Sites of Metastases at Start of Lorlatinib Treatment
Description: Number of participants according to sites of metastases at start of lorlatinib treatment were presented in this outcome measure. One participant could have more than one site of metastases.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Lorlatinib 2L | Lorlatinib 3L or Later
Number analyzed (Participants) | 29 | 22
Participants
  Ipsilateral lung | 11 | 7
  Contralateral lung | 7 | 5
  Lymph node affiliation | 23 | 18
  Remote lymph node | 5 | 6
  Liver | 7 | 4
  Bone | 17 | 14
  Brain | 13 | 12
  Adrenal glands | 1 | 2
  Kidney | 1 | 0
  Other | 11 | 5

15. Primary Outcome: Number of Participants According to Presence of Previous Medical History
Description: Number of participants with previous medical history related to history of treatment for ALK+ NSCLC were reported in this outcome measure.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Lorlatinib 2L | Lorlatinib 3L or Later
Number analyzed (Participants) | 29 | 22
Participants
  No | 17 | 15
  Yes | 12 | 7

16. Primary Outcome: Number of Participants According to Details of Previous Medical History
Description: Number of participants with previous medical history of high blood pressure, diabetes, hyperlipidemia and other were reported in this outcome measure.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Lorlatinib 2L | Lorlatinib 3L or Later
Number analyzed (Participants) | 12 | 7
Participants
  High blood pressure | 0 | 0
  Diabetes | 0 | 0
  Hyperlipidemia | 0 | 0
  Other | 12 | 7

17. Primary Outcome: Number of Participants According to Presence of Complications
Description: Complication was defined as a disease or disorder arising as a consequence of another disease. Number of participants according to presence of complications were reported in this outcome measure.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Lorlatinib 2L | Lorlatinib 3L or Later
Number analyzed (Participants) | 29 | 22
Participants
  No | 17 | 13
  Yes | 12 | 9

18. Primary Outcome: Number of Participants According to Details of Complications
Description: Number of participants who developed complications such as high blood pressure, diabetes, hyperlipidemia and other were reported in this outcome measure. One participant may have more than one complication.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Lorlatinib 2L | Lorlatinib 3L or Later
Number analyzed (Participants) | 12 | 9
Participants
  High blood pressure | 4 | 2
  Diabetes | 4 | 2
  Hyperlipidemia | 7 | 2
  Other | 9 | 7

19. Primary Outcome: Number of Participants According to Smoking History
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Lorlatinib 2L | Lorlatinib 3L or Later
Number analyzed (Participants) | 29 | 22
Participants
  Current | 7 | 5
  Former | 8 | 6
  Never | 14 | 11

20. Primary Outcome: Brinkman Index Score
Description: The Brinkman index (BI) is a measure of cigarette smoke exposure and is used as a predictor of chronic obstructive pulmonary disease (COPD) in smokers. It is calculated as the number of cigarettes smoked per day multiplied by the number of years of smoking. The scores ranged from 20 to 1050, where higher scores indicated higher cigarette smoke exposure.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: (Cigarettes per day)*years
Arm/Group | Lorlatinib 2L | Lorlatinib 3L or Later
Number analyzed (Participants) | 15 | 9
(Cigarettes per day)*years | 366.7 (271.1) | 262.9 (314.1)

21. Primary Outcome: Number of Participants With Anaplastic Lymphoma Kinase (ALK) Test Result
Description: ALK test was used to detect specific rearrangements in the ALK gene in cancer cells and tissue. Number of participants with ALK test result were reported in this outcome measure.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Lorlatinib 2L | Lorlatinib 3L or Later
Number analyzed (Participants) | 29 | 22
Participants | 29 | 22

22. Primary Outcome: Number of Participants According to Type of ALK Testing Method
Description: Number of participants according to the type of ALK testing methods including immunohistochemistry (IHC), fluorescence in situ hybridization (FISH), reverse transcription polymerase chain reaction (RT-PCR) and other methods were presented in this outcome measure. One participant may have more than one type of ALK testing method.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Lorlatinib 2L | Lorlatinib 3L or Later
Number analyzed (Participants) | 29 | 22
Participants
  IHC | 21 | 13
  FISH | 15 | 12
  RT-PCR | 2 | 4
  Other | 1 | 1

23. Primary Outcome: Number of Participants for Whom Dates of ALK Test Was Available
Description: Number of participants for whom dates of performing ALK test was available was presented in this outcome measure.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Lorlatinib 2L | Lorlatinib 3L or Later
Number analyzed (Participants) | 29 | 22
Participants | 29 | 22

24. Primary Outcome: Number of Participants According to Treatment Administered for NSCLC Prior to Start of Lorlatinib Treatment
Description: Number of participants according to treatment administered (Anaplastic Lymphoma Kinase- Tyrosine Kinase Inhibitor [ALK-TKI] including brigatinib, ceritinib and crizotinib or Other chemotherapy]) for NSCLC prior to start of lorlatinib treatment were presented in this outcome measure.
Time Frame: Prior to initiation of lorlatinib treatment (up to approximately 23.7 months); retrospective data was retrieved and analyzed during 4 months of this observational study
Population: FAS: participants with confirmed ALK+ NSCLC who started treatment with lorlatinib as second-line or later therapy from 01-May-2019 to 31-Dec-2020 and had confirmed treatment with alectinib in first line setting in a medical record. Only participants with any prior therapy for NSCLC other than alectinib as first line were analysed. All participants in Lorlatinib 2L arm were administered first line treatment of alectinib and did not receive any prior therapy for NSCLC other than alectinib.
Measure: Count of Participants; unit: Participants
Arm/Group | Lorlatinib 2L | Lorlatinib 3L or Later
Number analyzed (Participants) | 0 | 22
Participants
  ALK-TKI |  | 7
  Other chemotherapy |  | 15

25. Primary Outcome: Time to Treatment Failure for Lorlatinib as the Second Line Therapy and the Third or Later Line Therapy
Description: Time to treatment failure (TTF) was the time from the first date of lorlatinib treatment to the date of any-cause treatment discontinuation including disease progression, treatment toxicity and death. If participants continued treatment, TTF was censored at the available last date of treatment or the study end period. Disease progression (PD) was defined in a method that complied with Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 tumor assessment as closely as possible in clinical practice by investigator's judgement. TTF was analyzed using Kaplan-Meier method.
Time Frame: From the date of initiation of lorlatinib treatment to the date of any-cause treatment discontinuation or study end, from 01-May-2019 to 15-Oct-2021 (approximately 30 months); retrospective data was retrieved and analyzed during 4 months of this study
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lorlatinib 2L | Lorlatinib 3L or Later
Number analyzed (Participants) | 29 | 22
Months | 10.8 [3.9 to 13.8] | 11.5 [2.9 to NA] — Upper limit of 95% confidence interval was not estimable due to insufficient number of participants with events.

26. Secondary Outcome: Number of Participants According to Reasons for Discontinuation of Each Treatment Line of Therapy for Lorlatinib
Time Frame: From the date of initiation of lorlatinib treatment to the date of any-cause treatment discontinuation, from 01-May-2019 to 15-Oct-2021 (approximately 30 months); retrospective data was retrieved and analyzed during 4 months of this study
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Lorlatinib 2L | Lorlatinib 3L or Later
Number analyzed (Participants) | 20 | 14
Participants
  Progression disease | 16 | 9
  Adverse event | 3 | 4
  Other | 1 | 1

27. Secondary Outcome: Objective Response Rate for Lorlatinib as the Second Line Therapy and the Third Line or Later Therapy
Description: Objective response rate was defined as the percentage of participants with best overall response (BOR) of either complete response (CR) or partial response (PR) according to RECIST version 1.1 from first date lorlatinib treatment until date of treatment discontinuation. CR: disappearance of target and non-target lesions, with exception of nodal disease and normalization of tumor markers. All nodes, target and non-target must have short axis measures <10 mm. PR: >=30% decrease in sum of measures (longest diameter for tumor lesions and short axis measure for nodes) of target lesions, taking as reference baseline sum of diameters. Non-target lesions must be non-PD. PD was defined in a method that complied with RECIST version 1.1 tumor assessment as closely as possible in clinical practice by investigator's judgement.
Time Frame: From the date of initiation of lorlatinib treatment to the date of treatment discontinuation, from 01-May-2019 to 15-Oct-2021 (approximately 30 months); retrospective data was retrieved and analyzed during 4 months of this observational study
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Lorlatinib 2L | Lorlatinib 3L or Later
Number analyzed (Participants) | 29 | 22
Percentage of participants | 44 [24.4 to 65.1] | 23.5 [6.8 to 49.9]

28. Secondary Outcome: Time to Treatment Failure for Alectinib as the First-Line Therapy: Overall Participants
Description: Time to treatment failure was the time from the first date of alectinib treatment to the date of any-cause treatment discontinuation including disease progression, treatment toxicity and death. If participants continued treatment, TTF was censored at the available last date of treatment or the study end period. PD was defined in a method that complied with RECIST version 1.1 tumor assessment as closely as possible in clinical practice by investigator's judgement. TTF was analyzed using Kaplan-Meier method.
Time Frame: From the date of initiation of alectinib treatment to the date of any-cause treatment discontinuation or study end (maximum of 61.8 months of alectinib treatment); retrospective data was retrieved and analyzed during 4 months of this observational study
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Overall Participants: Participants with ALK+ NSCLC who started treatment with lorlatinib as the second-line or later line therapy from 01-May- 2019 to 31-Dec-2020 in clinical practice after failure of alectinib treatment as the first line therapy were included.
Arm/Group | Overall Participants
Number analyzed (Participants) | 51
Months | 18.1 [10.5 to 24.2]

29. Secondary Outcome: Time to Treatment Failure for Subsequent Other Treatment
Description: Time to treatment failure was the time from the first date of the other subsequent treatment to the date of other subsequent treatment discontinuation including disease progression, treatment toxicity and death. If participants continued treatment, TTF was censored at the available last date of treatment or the study end period. PD was defined in a method that complied with RECIST version 1.1 tumor assessment as closely as possible in clinical practice by investigator's judgement. TTF was analyzed using Kaplan-Meier method.
Time Frame: From the date of initiation of subsequent other treatment to the date of any-cause treatment discontinuation or study end (maximum of 22.9 months of subsequent other treatment); retrospective data was retrieved and analyzed during 4 months of this study
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lorlatinib 2L | Lorlatinib 3L or Later
Number analyzed (Participants) | 15 | 7
Months | NA [NA to NA] — Median, upper and lower limits of 95% CI could not be calculated due to insufficient number of participants with events | NA [NA to NA] — Median, upper and lower limits of 95% CI could not be calculated due to insufficient number of participants with events

30. Secondary Outcome: Objective Response Rate for Alectinib
Description: Objective response rate was defined as the percentage of participants with BOR of either CR or PR according to RECIST version 1.1 from the first date of alectinib until the date of treatment discontinuation. CR = disappearance of target and non-target lesions, with exception of nodal disease and normalization of tumor markers. All nodes, both target and non-target must have short axis measures <10 mm. PR = at least a 30% decrease in the sum of measures (longest diameter for tumor lesions and short axis measure for nodes) of target lesions, taking as reference baseline sum of diameters. Non-target lesions must be non-PD. PD was defined in a method that complied with RECIST version 1.1 tumor assessment as closely as possible in clinical practice by investigator's judgement.
Time Frame: From the date of initiation of alectinib treatment to the date of any-cause treatment discontinuation (maximum of 61.8 months of alectinib treatment); retrospective data was retrieved and analyzed during 4 months of this observational study
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Lorlatinib 2L | Lorlatinib 3L or Later
Number analyzed (Participants) | 29 | 22
Percentage of participants | 69.2 [48.2 to 85.7] | 94.7 [74.0 to 99.9]

31. Secondary Outcome: Combined Time to Treatment Failure of the Sum of Alectinib and Subsequent Therapy Including TTF of Lorlatinib as the Second Line Therapy and the Third Line or Later Therapy
Description: Combined TTF is defined as sum of the time from the first date of alectinib to the date of any-cause alectinib discontinuation, the time from the first date of lorlatinib to the date of lorlatinib discontinuation and the time from the first date of the other subsequent treatment to the date of other subsequent treatment discontinuation. If participants continued treatment, combined TTF was censored at the available last date of treatment or the study end period. Combined TTF was analyzed using Kaplan-Meier method.
Time Frame: From date of initiation of alectinib treatment until date of treatment discontinuation or study end, from Sep-2014 until 15-Oct-2021 (up to approximately 85 months); retrospective data was retrieved and analyzed during 4 months of this study
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lorlatinib 2L | Lorlatinib 3L or Later
Number analyzed (Participants) | 29 | 22
Months | NA [27.2 to NA] — Median and upper limit of 95% confidence interval was not estimable due to insufficient number of participants with events. | 55.0 [34.9 to NA] — Upper limit of 95% confidence interval was not estimable due to insufficient number of participants with events.

32. Secondary Outcome: Time to Last Treatment Failure for Lorlatinib as the Second Line Therapy and the Third Line or Later Therapy
Description: Time to last treatment failure (TLTF) is the time from the first date of lorlatinib to the date of any-cause treatment discontinuation including disease progression, treatment toxicity and death in the last treatment. If participants continued treatment, TLTF was censored at the available last date of treatment or the study end period. PD was defined as >= 20% increase in sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to relative increase of 20%, sum must also demonstrate an absolute increase of at least 5 mm and appearance of one or more new lesions. TLTF was analyzed using Kaplan-Meier method.
Time Frame: as for outcome 25
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lorlatinib 2L | Lorlatinib 3L or Later
Number analyzed (Participants) | 29 | 22
Months | NA [32.2 to NA] — Median and upper limit of 95% confidence interval was not estimable due to insufficient number of participants with events. | 59.7 [35.5 to NA] — Upper limit of 95% confidence interval was not estimable due to insufficient number of participants with events.

ADVERSE EVENTS:
Time Frame: Not applicable as adverse events were not collected during the study
Description: This observational retrospective study retrieved data from medical records and the data existed as unstructured data. In these data sources, individual participant data were not retrieved or validated, and it was not possible to link a particular product and medical event for any individual. Thus, the minimum criteria for reporting an adverse event could not be met, hence safety data were not collected and reported.
Arm/Group | Lorlatinib 2L | Lorlatinib 3L or Later
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-04-15): https://cdn.clinicaltrials.gov/large-docs/88/NCT04979988/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-12): https://cdn.clinicaltrials.gov/large-docs/88/NCT04979988/SAP_001.pdf